CLINICAL TRIAL: NCT06060964
Title: Enabling Remote Access to Breathe Easier: A Novel Approach to Improve Symptom Self-Management and Wellness for Survivors of Lung Cancer and Their Family Members
Brief Title: Enabling Remote Access to Breathe Easier: A Novel Approach to Improve Symptom Management
Acronym: Breathe Easier
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Otis (Shaun) Owens, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 00122553
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Lung Cancer, Nonsmall Cell; Lung Cancer Stage I; Lung Cancer Stage II; Lung Cancer Stage III
Keywords: mindfulness; lung cancer; technology
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this group will use the Breathe Easier progressive web application each day for a period of 8-weeks.
  Interventions: Other: Breathe Easier Progressive Web Application
- Non-intervention Group (Control Group) (No Intervention): Participants in this group will receive no intervention.

INTERVENTIONS:
Other: Breathe Easier Progressive Web Application — The Breathe Easier Progressive Web Application is an 8-week, mindfulness based cancer recovery training program consisting of breathing retraining exercises, mindfulness meditation, gentle yoga, and cancer-specific educational activities, guided by a combination of written instructions, video, and audio. The progressive web application can be downloaded onto any mobile device.
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to evaluate the preliminary affects of "Breathe Easier," an evidence-based multi-level mindfulness intervention (i.e., progressive web application) for survivors of lung cancer. The key aims of this study are to (1) Evaluate the feasibility (usability, acceptability intervention adherence) of the "Breathe Easier" and (2) assess the impact of the intervention on dyspnea, fatigue, and quality of life among survivors of lung cancer. Participants in the intervention group will use the "Breathe Easier" progressive web application for a period of 8-weeks, while participants in the control group will receive no intervention. Researchers will compare the intervention and control groups to see if there are salient differences in dyspnea, fatigue, and quality of life between the two groups.

DETAILED DESCRIPTION:
Cancer, a major health problem worldwide, is the second leading cause of death in the United States. As cancer death rates drop, the population of survivors of cancer is growing, projected to reach 18 million by 2022, with an estimated 800,000 of those being long-term survivors. Lung cancer is the second-most diagnosed cancer, accounting for more cancer deaths than breast, colorectal, and prostate cancers combined. Approximately 80% of patients with lung cancer will be diagnosed with non-small cell lung cancer (NSCLC), and about 25% will present with early-stage or localized disease (stages I-III). Lower prevalence of cigarette smoking, screening improvements, and treatment advances are improving five-year survival rates (currently 59% for stages I-II, 32% for stage III) [1-3]. Survivors of lung cancer will not only be more numerous but will be living longer. A diagnosis of lung cancer provides an opportunity to introduce targeted, effective, family-focused interventions. Developing interventions for self-managing lung cancer as a chronic illness is imperative. This project supports the strategic research priorities of the National Institute of Nursing Research (NINR) and National Cancer Institute (NCI) by developing and testing an evidence-based multi-level mindfulness intervention, Breathe Easier (BE), using the ORBIT model for behavioral intervention development and a theory-guided approach based on the individual and family self-management theory (IFSMT). BE empowers survivors and family members to manage symptoms and change unhealthy behaviors together.

SPECIFIC AIMS: The long-term goal of our research is to improve outcomes for survivors of NSCLC, stages I-III, and their family members. Our specific aims are as follows:

(1) Evaluate the feasibility (usability, acceptability intervention adherence) of BE and (2) Assess the preliminary effects (dyspnea, fatigue, quality of life) among survivors of lung cancer who receive the intervention as compared with those who do not receive BE.

ELIGIBILITY:
Inclusion Criteria:

* Must be a White or African-American survivor of NSCLC, stages I-III, have access to a smart phone, have internet access, and be willing and able to use a mobile application and participate in daily meditations/gentle movement exercises for 8-weeks.

Exclusion Criteria:

* Persons not meeting all inclusion criteria will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-10-02 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Fatigue (FACIT Fatigue Scale v. 4) | Administered prior to the start of intervention and immediately following the intervention.
  13 items measuring individual fatigue during usual activity level over the past 7 days; 4-point Likert scale, ranging from 4 (Not at All Fatigued) to 0 (Very Much Fatigued). Scores range 0-52 (< 30 indicates severe fatigue)
Dyspnea (MRC Breathlessness Scale) | Administered prior to the start of intervention and immediately following the intervention.
  1 item, comprised of five statements that describe almost the entire range of respiratory disability from none (Grade 1) to almost complete incapacity (Grade 5). It can be self-administered by asking subjects to choose a phrase that best describes their condition, e.g. 'I only get breathless with strenuous exertion' (Grade 1) or 'I am too breathless to leave the house' (Grade 5)
Quality of Life (SF-36 Medical Outcomes Survey) | Administered prior to the start of intervention and immediately following the intervention.
  36 items that are meant to reflect 8 domains of health, including physical functioning, physical role, pain, general health, vitality, social function, emotional role, and mental health. Likert scales and yes/no options are used to assess function and well-being on this 36-item questionnaire.

SECONDARY OUTCOMES:
Usability (System Usability Scale) | Administered only to intervention group immediately following the 8-week intervention
  10 items measuring usability; 5-point Likert scale, ranging from 1 (Strongly disagree) to 5 (Strongly disagree). Converted scores range from 0 to 100 (> 68 indicates average usability)
Acceptability (Acceptability of Intervention Measure) | Administered only to intervention group immediately following the 8-week intervention
  4-items measuring perceived intervention acceptability; 5-point Likert scale ranging from 1 (Completely Disagree) to 5 (Completely Agree). Score is creating by calculated mean across items.
Intervention Adherence | Administered only to intervention group immediately following the 8-week intervention
  number of intervention days/activities completed.

CONTACTS AND LOCATIONS:
Overall Officials: Otis Owens, PhD, Principal Investigator — Associate Professor; Karen McDonnell, PhD, Principal Investigator — Associate Professor
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
At this time, there is no plan to make individual participant data available.